CLINICAL TRIAL: NCT01481974
Title: An Evaluation of the Safety and Preliminary Efficacy of Perioperative Treprostinil in Preventing Ischemia and Reperfusion Injury in Adult Orthotopic Liver Transplant Recipients
Brief Title: Safety and Efficacy of Treprostinil in Ischemia and Reperfusion Injury in Adult Orthotopic Liver Transplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abhinav Humar, MD (Other)
Responsible Party: Sponsor-Investigator, Abhinav Humar, MD, MD, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19100094
Record Dates: First submitted 2011-10-20; First posted 2011-11-30 (Estimated); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Ischemia Reperfusion Injury
Keywords: liver transplantation; treprostinil
MeSH Terms: conditions — Reperfusion Injury | interventions — treprostinil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treprostinil (Experimental): This is a single center, open-label, dose-escalation Phase I/II study of Treprostinil.
  Interventions: Drug: Treprostinil

INTERVENTIONS:
Drug: Treprostinil — The Treatment Phase will begin at the initiation of Treprostinil after induction of anesthesia for the transplant surgery and continues throughout the surgery and for approximately a total of 120 hours.
  Treatment phase activities include:
  • Initiation of Treprostinil after the patient is hemodynamically stable following transplant surgery. (Treprostinil dosing will follow a standard 3 + 3 phase 1 design.
  Other Names: Brand name: REMODULIN

SUMMARY:
The overall purpose of this study is to evaluate the safety, pharmacokinetics and preliminary efficacy of a five-days post-operative course of Treprostinil in liver transplant patients.

The hypothesis of this study is that Treprostinil can be safely administered post-operatively in liver transplant patients. Once safety is documented future studies will address its ability to ameliorate or prevent reperfusion mediated dysfunction of the liver graft and thereby reduce morbidity, leading to shorter hospital stays as compared to historical controls.

DETAILED DESCRIPTION:
Prostaglandin-class drugs, including prostacyclin and its analogs, could represent an important advance toward the goal of reducing transplant related morbidity, mortality and associated costs by minimizing the effect of ischemia and re perfusion injury of the liver graft. Additionally, the reduction in serum creatinine and reduced need for post operative dialysis observed in some studies has implications in protecting the kidneys from the nephrotoxic affects of the immunosuppressant agents, especially during the early post-operative period. Routine use of prostaglandins (PGE1 and PGI2), however, was limited by its instability and short half life.

Treprostinil, as a prostanoid (prostacyclin analog), is expected to facilitate restoration of the blood supply to the revascularized graft and provide the well-characterized protective effects of this class of compounds in liver transplant patients. Treprostinil has the advantage of a longer elimination half-life than other prostanoids previously tested in these patients. Treprostinil is expected to significantly protect the graft from ischemia and re perfusion injury.

This is a pilot study to evaluate the safety, pharmacokinetics and preliminary efficacy of Treprostinil in orthotopic liver transplant patients as a first step to evaluate its use in prevention of ischemia and reperfusion injury of the grafted liver.

ELIGIBILITY:
Inclusion Criteria:

1. Have signed appropriate informed consent.
2. Be between 18 years and 65 years of age.
3. Have been accepted as a liver transplant candidate at the University of Pittsburgh Medical center (UPMC).
4. Be receiving a cadaver donor liver transplant.
5. Be treated in accordance with the standard of care protocol(s) currently in effect for liver transplant recipients at the UPMC, including immunosuppression and other elements of pre- and post-operative care.

Exclusion Criteria:

Subjects must not:

1. Be receiving a living donor liver transplant.
2. Be receiving a donor liver with a cold ischemia time less than 5 hours or greater than 12 hours.
3. Be receiving any investigational drug (a drug other than Treprostinil administered under an IND) or participating in any other investigational study, with the exception of alemtuzumab (Campath).
4. Be receiving any prostanoid to treat portopulmonary hypertension.
5. Have had a failed liver transplant within the previous 180 days.
6. Be undergoing multi-organ transplantation (transplantation of organs other than liver at the same time as the liver transplantation procedure).
7. Have fulminant hepatic failure
8. Model for end stage liver diseases (MELD) score of > 40
9. Hepatitis C positive donor liver
10. On renal replacement therapy at the time of study
11. Be receiving any non-standard immunosuppression protocol or other non-standard treatment that could affect interpretation of the study results.
12. Those currently receiving treatment for portopulmonary hypertension.
13. Those with significant cardiovascular disease including treatment with inotropes.
14. Have any known hypersensitivity to prostaglandins, prostacyclin or treprostinil.
15. If female, be pregnant or nursing (as confirmed by urine pregnancy test at Baseline).
16. HIV positive
17. Individuals who are allergic to iodine
18. Individuals who are receiving methylene blue
19. A donor liver with macrosteatosis greater than 40% if biopsy results are available

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2012-12; Primary Completion 2019-05-18 (Actual); Study Completion 2019-11-24 (Actual)

PRIMARY OUTCOMES:
Serum ALT concentration after treprostinil treatment in liver transplant patients | Day 7
  The liver injury marker such as alanine aminotransferase (ALT) will be measured in order to evaluate the protective effect of treprostinil in liver transplant recipients.

SECONDARY OUTCOMES:
Pharmacokinetics of treprostinil in liver transplant patients | 0, 2, 4, 6, 12, 18, 24, 30, 36, 42, 48, 72, 96 and 120 hrs during therapy and approximately 0.5, 1, 2, 4, 6, 8, 12 and 24 hr post study drug termination
  Clearance and half life

CONTACTS AND LOCATIONS:
Overall Officials: Abhinav Humar, M.D., Principal Investigator — University of Pittsburgh Medical Center
Locations (2):
- United States (2):
  - Abhinav Humar, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania